CLINICAL TRIAL: NCT00897676
Title: Role of GLP-1 in Congenital Hyperinsulinism:Effect of Exendin-(9-39) on Fasting Adaptation and Protein Sensitivity
Brief Title: Effect of Exendin-(9-39) on Fasting Adaptation and Protein Sensitivity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Diva De Leon (Other)
Responsible Party: Sponsor-Investigator, Diva De Leon, M.D. Assistant Professor of Pediatrics, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008-10-6255; R01FD004905 (Other Grant/Funding Number: US Food and Drug Administration)
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Congenital Hyperinsulinism
Keywords: Hyperinsulinism; Hypoglycemia; KATP channel
MeSH Terms: conditions — Congenital Hyperinsulinism; Hyperinsulinism; Hypoglycemia | interventions — exendin (9-39); Saline Solution

STUDY DESIGN:
Intervention Model Description: In a random crossover design, subjects were assigned to either intervention (6 hour infusion of exendin( 9-39) at a dose range of 100-500pmol/kg/min) or vehicle (6hr infusion of 0.9%NaCl)
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle first, then Exendin-(9-39) (Other): An infusion of vehicle (0.9%NaCl) will run for 60 minutes(time -60 to 0) before starting the study infusion of vehicle or exendin-(9-39). At time 0, vehicle (0.9%NaCl) will be started and will continue for 6 hours. The following day, at time 0, exendin-(9-39) at a dose ranging from 100-500pmol/kg/min will be started and continue for 6 hours. During both infusions, blood glucose, insulin, c-peptide, GLP-1, and glucagon will be measured every 30 minutes.
  Interventions: Drug: Exendin-(9-39); Drug: placebo
- Exendin-(9-39) first then Vehicle. (Other): An infusion of vehicle (0.9%NaCl) will run for 60 minutes(time -60 to 0) before starting the study infusion of vehicle or exendin-(9-39). . At time 0, exendin-(9-39) at a dose ranging from 100-500pmol/kg/min will be started and continue for 6 hours. The following day, at time 0, vehicle (0.9%NaCl) will be started and will continue for 6 hours. During both infusions, blood glucose, insulin, c-peptide, GLP-1, and glucagon will be measured every 30 minutes.
  .
  Interventions: Drug: Exendin-(9-39); Drug: placebo

INTERVENTIONS:
Drug: Exendin-(9-39) — 100-500pmol/kg/min
Drug: placebo — placebo (0.9% NaCl)
  Other Names: (0.9% NaCl)

SUMMARY:
The purpose of this study is to examine the effects of exendin-(9-39) on fasting blood glucose and protein induced hypoglycemia on subjects with Congenital Hyperinsulinism. Funding Source - FDA Office of Orphan Products Development (OODP).

DETAILED DESCRIPTION:
This is a placebo controlled study with randomized crossover design to evaluate the effect of the glucagon-like peptide-1 (GLP-1) receptor antagonist, exendin-(9-39), on fasting blood glucose levels, protein-induced hypoglycemia, and fasting tolerance of subjects with congenital hyperinsulinism due to mutations in the ATP- sensitive potassium channel (KATP) channel.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of hyperinsulinism
* Mutation analysis results demonstrating KATP channel defect
* Age 6 months to 18 years with
* Persistent hypoglycemia

Exclusion Criteria:

* Current therapy with medications that may affect glucose metabolism such as octreotide, diazoxide, high dose glucocorticoids, adrenergic agents, etc. Subjects will be eligible to participate if the last dose of octreotide is given 48 hrs before study day 1 and the last dose of diazoxide is given 72 hours before study day 1
* Evidence of a medical condition that might alter results or compromised the elimination of the peptide, including active infection, kidney failure, severe liver dysfunction, severe respiratory or cardiac failure
* Pregnancy
* Subjects with milk protein allergy will be excluded for participating in studies involving protein tolerance test

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2009-05; Primary Completion 2016-08-26 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diva D DeLeon, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stefanovski D, Vajravelu ME, Givler S, De Leon DD. Exendin-(9-39) Effects on Glucose and Insulin in Children With Congenital Hyperinsulinism During Fasting and During a Meal and a Protein Challenge. Diabetes Care. 2022 Jun 2;45(6):1381-1390. doi: 10.2337/dc21-2009. PMID 35416981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects age 6months to 18 years with congenital hyperinsulinism due to mutations in the Katp channel( KatpHI) were recruited from the Hyperinsulinism Center at The Children's Hospital of Philadelphia
Pre-assignment Details: 17 subject were enrolled (consented). One(1) withdrawn
Groups:
- Vehicle First Then Exendin-(9-39): An infusion of vehicle (0.9%NaCl) will run for 60 minutes(time -60 to 0) before starting the study infusion of vehicle or exendin-(9-39). At time 0, vehicle (0.9%NaCl) will be started and will continue for 6 hours. The following day, at time 0, exendin-(9-39) at a dose ranging from 100-500pmol/kg/min will be started and continue for 6 hours. During both infusions, blood glucose, insulin, c-peptide, glucagon-like peptide-(GLP-1) , and glucagon will be measured every 30 minutes.
  Vehicle: (0.9% NaCl)
- Exendin-(9-39) First Then Vehicle: An infusion of vehicle (0.9%NaCl) will run for 60 minutes(time -60 to 0) before starting the study infusion of vehicle or exendin-(9-39). At time 0, exendin-(9-39) at a dose ranging from 100-500pmol/kg/min will be started and continue for 6 hours. The following day, at time 0, vehicle (0.9%NaCl) will be started and will continue for 6 hours. During both infusions, blood glucose, insulin, c-peptide, glucagon-like peptide-(GLP-1) , and glucagon will be measured every 30 minutes.
  Exendin-(9-39): 100-500pmol/kg/min
Period: Intervention 1(6 Hours)
Arm/Group | Vehicle First Then Exendin-(9-39) | Exendin-(9-39) First Then Vehicle
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0
Period: Intervention 2(6 Hours)
Arm/Group | Vehicle First Then Exendin-(9-39) | Exendin-(9-39) First Then Vehicle
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subject Population: 9 subjects were randomized to the vehicle first arm and the next day they were switched to exendin- (9-39). 7 subjects were randomized to the exendin-(9-39) first arm and the next day they were switched to vehicle. All subjects enrolled and treated in the protocol served as their own control. Because of this and the small sample size, baseline characteristic data is presented together.
Arm/Group | Subject Population
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) Plasma Glucose
Description: Area under the curve plasma glucose from the initiation of infusion of vehicle or exendin-(9-39) to end of the infusion
Time Frame: Time 0 min - time 360 min
Population: A total of 16 subjects were included in the analysis. 1 subject was withdrawn.
Measure: Mean (Standard Deviation); unit: mg*min/dL
Groups:
- Vehicle: Subjects received an infusion of vehicle( 0.9%NaCl) intravenously from time 0 min to 360 min
  Vehicle: (0.9% NaCl)
- Exendin-(9-39): Subjects received an infusion of exendin-(9-39) intravenously at a dose ranging from 100-500pmol/kg/min from time 0 min to 360 min
  Exendin-(9-39)
Arm/Group | Vehicle | Exendin-(9-39)
Number analyzed (Participants) | 16 | 16
mg*min/dL | 26994.7 (4219.8) | 32122.2 (6650.1)

2. Secondary Outcome: Area Under the Curve (AUC) Plasma Insulin
Description: Area under the curve plasma insulin from the initiation of infusion of vehicle or exendin-(9-39) to end of the infusion
Time Frame: time 0 min to time 360 min
Population: data from only 15 subjects because the values were below the level of detection for one subject.
Measure: Mean (Standard Deviation); unit: uIU*min/mL
Groups:
- Vehicle: Subjects received an infusion of vehicle( 0.9%NaCl) intravenously from time 0 to time 360 min
  Vehicle: (0.9% NaCl)
- Exendin-(9-39): Subjects received an infusion of exendin-(9-39) intravenously from time 0 to time 360 min at a dose of 100-500 pmol/kg/min
  Exendin-(9-39)
Arm/Group | Vehicle | Exendin-(9-39)
Number analyzed (Participants) | 15 | 15
uIU*min/mL | 1578.7 (1089.9) | 1284.5 (553.7)

3. Secondary Outcome: Area Under the Curve (AUC) Plasma C-peptide
Description: Area under the curve plasma C-peptide from the beginning of the infusion of vehicle or exendin-(9-39) to the end of the infusion
Time Frame: time 0 min to time 360 min
Measure: Mean (Standard Deviation); unit: ng*min/mL
Groups:
- Vehicle: Subjects received an infusion of vehicle( 0.9%NaCl) intravenously from time 0 min to time 360 min
  Vehicle: (0.9% NaCl)
- Exendin-(9-39): Subjects received an infusion of exendin-(9-39) intravenously at a dose ranging from 100-500pmol/kg/min from time 0 min to time 360 min
  Exendin-(9-39)
Arm/Group | Vehicle | Exendin-(9-39)
Number analyzed (Participants) | 16 | 16
ng*min/mL | 281.4 (155.8) | 236.6 (112.5)

4. Secondary Outcome: Area Under the Curve (AUC) Plasma Glucagon
Description: Area under the curve plasma glucagon from the beginning of the infusion of vehicle or exendin-(9-39) to the end of the infusion
Time Frame: time 0 min to time 360 min
Measure: Mean (Standard Deviation); unit: pg*min/mL
Groups:
- Vehicle: Subjects receive an infusion of vehicle( 0.9%NaCl) intravenously from time 0 to time 360 min
  Vehicle: (0.9% NaCl)
- Exendin-(9-39): Subjects received an infusion of exendin-(9-39) intravenously at a dose ranging from 100-500pmol/kg/min from time 0 to time 360 min
  Exendin-(9-39)
Arm/Group | Vehicle | Exendin-(9-39)
Number analyzed (Participants) | 16 | 16
pg*min/mL | 22806.8 (10210.3) | 23409.4 (11396.1)

5. Secondary Outcome: Area Under the Curve ( AUC) Plasma Total GLP-1 (Glucagon-like Peptide-1)
Description: Area under the curve plasma total GLP-1 (glucagon-like peptide-1) from the beginning of the infusion of vehicle or exendin-(9-39) to the end of the infusion
Time Frame: time 0 to time 360 min
Measure: Mean (Standard Deviation); unit: pmol*min/L
Arm/Group | Vehicle | Exendin-(9-39)
Number analyzed (Participants) | 16 | 16
pmol*min/L | 4899.3 (2598.8) | 5698.8 (3484.8)

6. Secondary Outcome: Area Under the Curve ( AUC) Plasma Active GLP-1 (Glucagon-like Peptide-1)
Description: Area under the curve plasma active GLP-1 (glucagon-like peptide-1) from the beginning of the infusion of vehicle or exendin-(9-39) to the end of the infusion
Time Frame: time 0 min to time 360 min
Measure: Mean (Standard Deviation); unit: pmol*min/L
Groups:
- Vehicle: Subjects received an infusion of vehicle( 0.9%NaCl) intravenously from time 0 min to time 360 min
  Vehicle
Arm/Group | Vehicle | Exendin-(9-39)
Number analyzed (Participants) | 16 | 16
pmol*min/L | 1373.7 (1044) | 1432.9 (1114.3)

ADVERSE EVENTS:
Time Frame: baseline to 24 hours after the end of study of infusion.
Groups:
- Vehicle: Subjects received an infusion of vehicle (0.9% NaCl) intravenously from time 0 min to time 360 min
  Vehicle: (0.9% NaCl)
Arm/Group | Vehicle | Exendin-(9-39)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 12/16 | 8/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=16) | Exendin-(9-39) (N=16)
hypoglycemia (Endocrine disorders) | 11 (11) | 7 (7)
hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
For safety reasons, blood glucose levels were maintained above a safety threshold (55-60mg/dL) during the study by infusing dextrose intravenously which may limit the magnitude of the effect that we will be able to detect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes